CLINICAL TRIAL: NCT02449577
Title: Metabolomics in Beer Research: Identification of Biomarkers for Acute Intake of Beer and Alcohol in Individuals With a High or Low Habitual Intake, and Acute Effects on Plasma Glucose and Insulin Response Compared to Regular Soda
Brief Title: Identification of Biomarkers for Acute Intake of Beer and Alcohol and Acute Effects on Plasma and Insulin Response
Acronym: METABEER
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Carlsberg Breweries A/S (Unknown)
Responsible Party: Principal Investigator, Professor Lars Ove Dragsted, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: M212
Record Dates: First submitted 2013-06-28; First posted 2015-05-20 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Alcohol Consumption; Insulin Resistance
Keywords: Metabolomics; Beer; Biomarker; Glucose response; Insulin response
MeSH Terms: conditions — Alcohol Drinking; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (11):
- Beverage sequence ABCD (Experimental): Each participant randomized to this arm is exposed to 4 test meals in the order ABCD with a washout period of at least a week between each meal. Each meal consisted of a standardized lunch of Parisian toast (sandwichbread, ham, cheese) together with a beverage. Each beverage is assigned a letter, A, B, C, or D. The letter assignment is blinded. The following four drinks were used Placebo: 330 ml of a soft drink (Sports drink), Beer 1 - 330 ml of an alcohol-free beer (<0.1% alcohol), Beer 2 - 330 ml of a regular lager beer (4.6% alcohol), and Beer 3 - 330 ml of a strong beer (7.2% alcohol)
  Interventions: Other: Beverage sequence ABCD
- Beverage sequence CADB (Experimental): Each participant randomized to this arm is exposed to 4 test meals in the order CADB with a washout period of at least a week between each meal. Each meal consisted of a standardized lunch of Parisian toast (sandwichbread, ham, cheese) together with a beverage. Each beverage is assigned a letter, A, B, C, or D. The letter assignment is blinded. The following four drinks were used Placebo: 330 ml of a soft drink (Sports drink), Beer 1 - 330 ml of an alcohol-free beer (<0.1% alcohol), Beer 2 - 330 ml of a regular lager beer (4.6% alcohol), and Beer 3 - 330 ml of a strong beer (7.2% alcohol)
  Interventions: Other: Beverage sequence CADB
- Beverage sequence DACB (Experimental): Each participant randomized to this arm is exposed to 4 test meals in the order DACB with a washout period of at least a week between each meal. Each meal consisted of a standardized lunch of Parisian toast (sandwichbread, ham, cheese) together with a beverage. Each beverage is assigned a letter, A, B, C, or D. The letter assignment is blinded. The following four drinks were used Placebo: 330 ml of a soft drink (Sports drink), Beer 1 - 330 ml of an alcohol-free beer (<0.1% alcohol), Beer 2 - 330 ml of a regular lager beer (4.6% alcohol), and Beer 3 - 330 ml of a strong beer (7.2% alcohol)
  Interventions: Other: Beverage sequence DACB
- Beverage sequence CBAD (Experimental): Each participant randomized to this arm is exposed to 4 test meals in the order CBAD with a washout period of at least a week between each meal. Each meal consisted of a standardized lunch of Parisian toast (sandwichbread, ham, cheese) together with a beverage. Each beverage is assigned a letter, A, B, C, or D. The letter assignment is blinded. The following four drinks were used Placebo: 330 ml of a soft drink (Sports drink), Beer 1 - 330 ml of an alcohol-free beer (<0.1% alcohol), Beer 2 - 330 ml of a regular lager beer (4.6% alcohol), and Beer 3 - 330 ml of a strong beer (7.2% alcohol)
  Interventions: Other: Beverage sequence CBAD
- Beverage sequence ABDC (Experimental): Each participant randomized to this arm is exposed to 4 test meals in the order ABDC with a washout period of at least a week between each meal. Each meal consisted of a standardized lunch of Parisian toast (sandwichbread, ham, cheese) together with a beverage. Each beverage is assigned a letter, A, B, C, or D. The letter assignment is blinded. The following four drinks were used Placebo: 330 ml of a soft drink (Sports drink), Beer 1 - 330 ml of an alcohol-free beer (<0.1% alcohol), Beer 2 - 330 ml of a regular lager beer (4.6% alcohol), and Beer 3 - 330 ml of a strong beer (7.2% alcohol)
  Interventions: Other: Beverage sequence ABDC
- Beverage sequence DABC (Experimental): Each participant randomized to this arm is exposed to 4 test meals in the order DABC with a washout period of at least a week between each meal. Each meal consisted of a standardized lunch of Parisian toast (sandwichbread, ham, cheese) together with a beverage. Each beverage is assigned a letter, A, B, C, or D. The letter assignment is blinded. The following four drinks were used Placebo: 330 ml of a soft drink (Sports drink), Beer 1 - 330 ml of an alcohol-free beer (<0.1% alcohol), Beer 2 - 330 ml of a regular lager beer (4.6% alcohol), and Beer 3 - 330 ml of a strong beer (7.2% alcohol)
  Interventions: Other: Beverage sequence DABC
- Beverage sequence DCAB (Experimental): Each participant randomized to this arm is exposed to 4 test meals in the order DCAB with a washout period of at least a week between each meal. Each meal consisted of a standardized lunch of Parisian toast (sandwichbread, ham, cheese) together with a beverage. Each beverage is assigned a letter, A, B, C, or D. The letter assignment is blinded. The following four drinks were used Placebo: 330 ml of a soft drink (Sports drink), Beer 1 - 330 ml of an alcohol-free beer (<0.1% alcohol), Beer 2 - 330 ml of a regular lager beer (4.6% alcohol), and Beer 3 - 330 ml of a strong beer (7.2% alcohol)
  Interventions: Other: Beverage sequence DCAB
- Beverage sequence DBCA (Experimental): Each participant randomized to this arm is exposed to 4 test meals in the order DBCA with a washout period of at least a week between each meal. Each meal consisted of a standardized lunch of Parisian toast (sandwichbread, ham, cheese) together with a beverage. Each beverage is assigned a letter, A, B, C, or D. The letter assignment is blinded. The following four drinks were used Placebo: 330 ml of a soft drink (Sports drink), Beer 1 - 330 ml of an alcohol-free beer (<0.1% alcohol), Beer 2 - 330 ml of a regular lager beer (4.6% alcohol), and Beer 3 - 330 ml of a strong beer (7.2% alcohol)
  Interventions: Other: Beverage sequence DBCA
- Beverage sequence ADCB (Experimental): Each participant randomized to this arm is exposed to 4 test meals in the order ADCB with a washout period of at least a week between each meal. Each meal consisted of a standardized lunch of Parisian toast (sandwichbread, ham, cheese) together with a beverage. Each beverage is assigned a letter, A, B, C, or D. The letter assignment is blinded. The following four drinks were used Placebo: 330 ml of a soft drink (Sports drink), Beer 1 - 330 ml of an alcohol-free beer (<0.1% alcohol), Beer 2 - 330 ml of a regular lager beer (4.6% alcohol), and Beer 3 - 330 ml of a strong beer (7.2% alcohol)
  Interventions: Other: Beverage sequence ADCB
- Beverage sequence BADC (Experimental): Each participant randomized to this arm is exposed to 4 test meals in the order BADC with a washout period of at least a week between each meal. Each meal consisted of a standardized lunch of Parisian toast (sandwichbread, ham, cheese) together with a beverage. Each beverage is assigned a letter, A, B, C, or D. The letter assignment is blinded. The following four drinks were used Placebo: 330 ml of a soft drink (Sports drink), Beer 1 - 330 ml of an alcohol-free beer (<0.1% alcohol), Beer 2 - 330 ml of a regular lager beer (4.6% alcohol), and Beer 3 - 330 ml of a strong beer (7.2% alcohol)
  Interventions: Other: Beverage sequence BADC
- Beverage sequence ACDB (Experimental): Each participant randomized to this arm is exposed to 4 test meals in the order ACDB with a washout period of at least a week between each meal. Each meal consisted of a standardized lunch of Parisian toast (sandwichbread, ham, cheese) together with a beverage. Each beverage is assigned a letter, A, B, C, or D. The letter assignment is blinded. The following four drinks were used Placebo: 330 ml of a soft drink (Sports drink), Beer 1 - 330 ml of an alcohol-free beer (<0.1% alcohol), Beer 2 - 330 ml of a regular lager beer (4.6% alcohol), and Beer 3 - 330 ml of a strong beer (7.2% alcohol)
  Interventions: Other: Beverage sequence ACDB

INTERVENTIONS:
Other: Beverage sequence ABCD — Participants receive test beverages in the randomised order ABCD
  Arms: Beverage sequence ABCD
Other: Beverage sequence CADB — Participants receive test beverages in the randomised order CADB
  Arms: Beverage sequence CADB
Other: Beverage sequence DACB — Participants receive test beverages in the randomised order DACB
  Arms: Beverage sequence DACB
Other: Beverage sequence CBAD — Participants receive test beverages in the randomised order CBAD
  Arms: Beverage sequence CBAD
Other: Beverage sequence ABDC — Participants receive test beverages in the randomised order ABDC
  Arms: Beverage sequence ABDC
Other: Beverage sequence DABC — Participants receive test beverages in the randomised order DABC
  Arms: Beverage sequence DABC
Other: Beverage sequence DCAB — Participants receive test beverages in the randomised order DCAB
  Arms: Beverage sequence DCAB
Other: Beverage sequence DBCA — Participants receive test beverages in the randomised order BDCA
  Arms: Beverage sequence DBCA
Other: Beverage sequence ADCB — Participants receive test beverages in the randomised order ADCB
  Arms: Beverage sequence ADCB
Other: Beverage sequence BADC — Participants receive test beverages in the randomised order BADC
  Arms: Beverage sequence BADC
Other: Beverage sequence ACDB — Participants receive test beverages in the randomised order ACDB
  Arms: Beverage sequence ACDB

SUMMARY:
The objective of the study is to identify biomarkers for acute intake of beer and alcohol in individuals with a high or low habitual intake. Furthermore, we wish to identify compounds and metabolites in different types of beer and alcohol, which can serve as compliance markers for intake under the test conditions (blood tests and urine samples). We also wish to determine the acute effects of these beverages on plasma glucose and insulin response, compared to regular soda.

DETAILED DESCRIPTION:
The study is designed as a randomized, 4-way single-blinded cross-over intervention study. The participants are randomized individually to the order by which they shall receive 4 test meals. There will be implemented a standardized lunch which includes respectively 1) Light/alcohol-free (Tuborg Super Light 0,1% alcohol), 2) Regular lager (4,6% alcohol), 3) Strong beer(7,2% alcohol) and 4) a control drink without alcohol but with the same energy content (carbohydrate and protein) as the average of the other beverages ("sportsdrink"). Besides 330 ml of each test drink, each test meal consists of grilled cheese sandwiches (Tulip Food Company) and the amount of toast adjusted according to the type of drink served with each meal, so the content of macronutrients is the same in each meal.

The study includes 16-20 participants, randomized as to which order they will receive the 4 test meals with a washout period of at least 6 days in between test days. Upon arrival the test persons are asked to urinate (baseline sample), and at the 1st visit they are then weighed, height is measured and body composition (bioimpedance) is measured. After resting briefly, a baseline blood sample is taken and blood pressure is measured (1st and 4th visit). 45 minutes after start of the test meal the first postprandial blood sample is taken, and again after 45, 120 and 180 minutes. Urine is collected again at 0-90 min, 90-180 min and 3-24 hours after the test meal. Participants are provided with containers and equipment for this purpose, and must submit samples on an ongoing basis to the Dept. of Nutrition, Exercise and Sports.

ELIGIBILITY:
Inclusion Criteria:

* Healthy man or woman in the age group 18-60 years
* Likes and tolerates pasta, tomatoes and cheese, and is not a vegetarian or vegan, since meat (beef and pork) is included in the standardized dinner, breakfast and in the test meal
* Habitual alcohol intake (high: up to 7/14 units per week for women/men) or low: 0-2 units per week for both genders
* Tolerates alcohol

Exclusion Criteria:

* Systematic infections, psychiatric conditions and metabolic disease, and any clinical condition and other condition/situation, which according to the experimenter's assessment makes the person unfit to participate in the study
* Donation of a larger amount of blood (more than 24 ml) e.g. in connection with donation or other scientific research study, during the study and 3 months before start of the study
* Alcohol intake above the Danish Health and Medicines Authority's recommended 7 respective 14 drinks (units) per week for women and men
* Have or have had a drug addiction
* Allergy or intolerance to any of the tested drinks, or to any other foods included in the study. The participant will be specifically screened for possible alcohol allergy or intolerance
* Nursing, pregnancy or planned pregnancy.
* Not capable of complying with the procedures stipulated in the protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) for glucose | 0-180 minutes
  Glucose is measured at 0, 45, 90, 120, and 180 min after the test meal and the area is determined by the trapezoid method.

SECONDARY OUTCOMES:
Area under the curve for insulin | 0-180 min
  Insulin is measured at 0, 45, 90, 120, and 180 min after the test meal and the area is determined by the trapezoid method.
Plasma concentration of fatty acid ethyl esters (FAEE) | Change from 0-180min
  Change in FAEE from baseline to 180min by LC-MS/MS analysis of plasma.
Blood level of ethanol | 180 min
  The amount of ethanol is measured via a breath test using an alcoholmeter.
Plasma beer metabolites (metabolic profiling with NMR and mass spectrometry). | After the intervention
  Explorative marker to identify new beer intake-related metabolites in plasma.
Urinary content of paraaminobenzoic acid (PABA) | 24hour pooled urine from each volunteer
  Total PABA metabolites by colorimetric assay to account for completeness of urine collection.
Urinary content of ethyl glucuronide (EtG) and ethyl sulphate (EtS) | 0-24 hours
  EtG and EtS by quantitative LC-MS/MS
Blood content of ethyl glucuronide (EtG) and ethyl sulphate (EtS) | 0-180 min
  EtG and EtS are measured at 0, 45, 90, 120 and 180 minutes and the difference between treatments is determined by multivariate ANOVA followed (if significantly different) by t-tests for each time point.
Urinary content of acetaldehyde (ethanal) | 0 -24 hrs
  Ethanal is measured by a kit and compared between treatments.
Urinary compounds of beer metabolites | 0-24 hrs
  Metabolic profiling of urine by NMR and mass spectrometry.
Blood pressure | baseline and at time -30min on the last day of intervention.
  Measurement of supine systolic and diastolic blood pressure
Body fat mass and body fat percentage | baseline
  Measurement of body fat mass and fat percentage by bioimpedance
Urinary creatinine | 0-24hrs
  Creatinine is measured by standard clinical chemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Lars O. Dragsted, Professor, Principal Investigator — Department of Nutrition, Exercise and Sports, University of Copenhagen, Rolighedsvej 30, 1958 Frederiksberg C, Denmark
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen, Frederiksberg C, Denmark